CLINICAL TRIAL: NCT05303467
Title: FRONTIER: A Feasibility Study to Evaluate the Safety of the TheRaSphere GliOblastoma (GBM) Device iN PaTIEnts With Recurrent GBM
Brief Title: A Feasibility Study to Evaluate the Safety of the TheraSphere Glioblastoma (GBM) Device in Patients With Recurrent GBM
Acronym: FRONTIER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2478
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The TheraSphere GBM Y-90 Glass Microsphere System (TheraSphere GBM) is an yttrium-90 (Y-90) glass microsphere therapy for selective internal radiation therapy (endovascular radiotherapy) in recurrent GBM patients. Groups A, B, and C will be enrolled concurrently. Up to 26 subjects will be enrolled in Groups A and C. Four subjects will be enrolled in Group B. Up to 6 subjects will be enrolled in Group D.
  Enrollment in Group D will not begin until the FDA approves an IDE supplement including all data through the primary safety endpoint from the four Group B subjects, as well as any available data from the Group A and C subjects at the time of submission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Treatment Group A (Experimental): Subjects in which the perfused volume encompasses the non-dominant hemisphere and non-eloquent regions of the brain. The projected radiation absorbed dose to the treatment volume is 40 Gy ±10%.
  Interventions: Device: TheraSphere GBM
- Treatment Group B (Experimental): Subjects in which the perfused volume encompasses the non-dominant hemisphere and eloquent regions of the brain. The projected radiation absorbed dose to the treatment volume is 40 Gy ±10%.
  Interventions: Device: TheraSphere GBM
- Treatment Group C (Experimental): Subjects in which the perfused volume encompasses the dominant hemisphere and non-eloquent regions of the brain. The projected radiation absorbed dose to the treatment volume is 40 Gy ±10%.
  Interventions: Device: TheraSphere GBM
- Treatment Group D (Experimental): Subjects in which the perfused volume encompasses the dominant hemisphere and eloquent regions of the brain. The projected radiation absorbed dose to the treatment volume is 40 Gy ±10%.
  Interventions: Device: TheraSphere GBM

INTERVENTIONS:
Device: TheraSphere GBM — Single treatment of TheraSphere GBM device
  Other Names: TheraSphere™ GBM Y-90 Glass Microspheres (TheraSphere GBM)

SUMMARY:
The FRONTIER Study is a prospective, interventional, single-arm, multi-center, study to assess the safety and technical feasibility of TheraSphere GBM in patients with recurrent GBM.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is a highly aggressive brain cancer with a grave prognosis, resulting in <7% of patients surviving to five years post-diagnosis. External beam radiotherapy (EBRT) is currently a mainstay treatment for GBM; however, the dose delivered is limited by side effects. The targeted radiotherapy of the TheraSphere GBM Y-90 Glass Microsphere System (TheraSphere GBM) has promising potential to provide GBM patients with reduced side effects compared to external beam radiotherapy as well as a more effective treatment for this catastrophic disease.

The TheraSphere GBM device utilized in the FRONTIER trial is an yttrium-90 (Y-90) glass microsphere therapy for selective internal radiation therapy (endovascular radiotherapy) in recurrent GBM patients. The TheraSphere GBM treatment utilizes intra-arterial delivery and takes advantage of blood flow and direct tumor delivery. Treatment can be delivered by specific placement of a catheter close to the tumor through known angiographic techniques currently utilized by neuro-endovascular or interventional radiology physicians. Angiographic evaluation prior to treatment allows identification of tumor feeding arteries and definition of the treatment volume. TheraSphere GBM could achieve a high tumor response rate based on delivery of a tumor absorbed dose that is not currently possible with EBRT.

In consideration of the potential benefit of a more localized, targeted treatment with a reduced side effect profile compared to other treatment options, and the potential impact on patients' quality of life for this devastating disease, this First-in-Human Early Feasibility Study (EFS) of the TheraSphere GBM Y-90 Glass Microsphere System for the treatment of recurrent GBM is being conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older and has signed and dated the trial informed consent form (ICF)
2. Life expectancy ≥ 12 weeks
3. Subject is willing and able to comply with the trial testing, procedures, and follow-up schedule
4. History of a histologically confirmed diagnosis of glioblastoma per 2021 WHO criteria
5. Have radiographic evidence of tumor progression/recurrence with measurable disease (≥ 1 cm to ≤ 5cm bidirectional diameters) by contrast-enhancement on MRI, according to RANO criteria
6. Prior surgery and treatment with combination of radiotherapy and chemotherapy ± Tumor Treating Fields (Optune®)
7. Prior cranial radiation dose < 66 Gy
8. WHO performance status ≤ 2
9. The interval since completion of cranial radiotherapy must be > 6 months, unless there is tissue confirmation of tumor recurrence/progression outside the previous radiation treatment field, in which case the interval since completion of cranial radiation must be at least 12 weeks
10. Interval since last systemic therapy until presumed date of intervention ≥ 1 cycle or ≥ 2 biological half-lives, i.e.

    1. ≥ 4 weeks since last dose of temozolomide
    2. ≥ 6 weeks since last dose of lomustine or other nitrosourea
    3. ≥ 2 weeks since last dose of a small molecule targeted agent (Tyrosine Kinase Inhibitor or similar)
    4. ≥ 6 weeks from last dose of last intravenous bevacizumab infusion, or other antibody-based VEGF therapy
11. If receiving steroids, patient should be on a stable or decreasing dose equivalent to dexamethasone ≤ 6 mg/d, for at least 7 days prior to registration
12. Have adequate organ and bone marrow function within 14 days prior to registration, as defined below:

    1. INR ≤ 1.2 (in absence of anticoagulation)
    2. Platelets ≥ 100,000/L
    3. Creatinine ≤1.5 mg/dL
    4. Absolute Neutrophil Count ≥1.5 x 10^9/L
    5. Hemoglobin ≥9.0 g/dL
13. Have a negative pregnancy test within 14 days prior to registration on study (for FOCBP, female of child-bearing potential)
14. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active must be using, or agree to use, a medically acceptable method of birth control as confirmed by the investigator
15. Angiographic Mapping Inclusion Criteria:

    1. Accessible neurovascular anatomy that allows for safe microcatheter placement (up to two locations) to infuse TheraSphere GBM to treat all of the T1 enhancing component of target lesion confirmed by neuro-interventional team.
    2. Total treatment volume is ≤ 150cc as determined by multidisciplinary team.
16. Additional Inclusion Criteria:

    1. Group A: perfused volume encompasses the non-dominant hemisphere and non-eloquent regions of the brain
    2. Group B: perfused volume encompasses the non-dominant hemisphere and eloquent regions of the brain
    3. Group C: perfused volume encompasses the dominant hemisphere and non-eloquent regions of the brain
    4. Group D: perfused volume encompasses the dominant hemisphere and eloquent regions of the brain

Exclusion Criteria:

1. Have bilateral gadolinium enhancing disease, tumor located in the posterior fossa, tumor involving critical subcortical structures (thalamus/hypothalamus, midbrain, brainstem, corticospinal tract, internal capsule, cerebral peduncle), tumor approximating or invading the brainstem and/or optic chiasma, leptomeningeal disease, or extracranial metastatic disease
2. Have received more than 1 course of prior cranial radiotherapy (EBRT)
3. Have received radiosurgery, brachytherapy, or hypofractionated radiotherapy
4. Have received more than 2 systemic treatment protocols (lines of treatment), not including maintenance temozolomide
5. Have received prior intra-arterial cerebral infusion therapy
6. Have received more than 2 surgical GBM-related procedures
7. Have received prior thoracic radiation therapy
8. Are at increased risk of wound dehiscence by the discretion of the investigators (e.g. brain surgery within the last 3 months, poor skin condition, and/or previously infected surgical field or any other condition that is of increased infectious risk in the opinion of the neurosurgeon)
9. Have uncontrolled epilepsy
10. Have severe and/or insufficiently controlled intercurrent illness; patients with the following are not eligible:

    1. Hypertension grade 3 or higher without adequate control on medications
    2. Symptomatic or unstable cardiac disease, known to have right-to-left shunts, or severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg)
    3. Pulmonary insufficiency (arterial oxygen pressure (Pa,O2) of < 60 mmHg, or oxygen saturation (Sa,O2) of < 90%) as measured by fingertip pulse oximeter
    4. Ongoing or active bacterial or viral infection requiring systemic treatment (including HIV)
    5. Pneumonitis
    6. Psychiatric illness/social situations that would limit compliance with study requirements
    7. Peripheral Neuropathy ≥ grade 1
    8. Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety, study endpoints or longevity
11. Are currently pregnant or breast feeding (unless patient agrees to stop breastfeeding)
12. Patients with a history of an active other malignancy within 1 year prior to registration. NOTE: Exceptions to this requirement include adequately treated non-melanoma skin cancer or lentigo maligna or carcinoma in situ without evidence of disease, or recurrent glioblastoma
13. Patients with a history of ischemic cerebral disease and/or at risk of cerebral herniation
14. Medical contraindication to undergo contrast-enhanced magnetic resonance imaging (MRI)
15. Known history of hypersensitivity reactions to iodinated and/or gadolinium-based contrast
16. Subject has received any other investigational agents within 4 weeks of treatment, or is currently participating, or plans to participate in, another investigational trial that may confound the results of this trial (unless written approval is received from the Boston Scientific study team)
17. Angiographic Mapping Exclusion Criteria: Patients with significant vascular disease, significant AV shunting, or anatomic tortuosity on MR/CT Angiogram precluding safe or feasible vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The number of grade 3-5 non-hematological toxicities | 30 days post index procedure
The number of ≥ grade 3 CNS toxicities related to non-target embolization | 30 days post index procedure
Occurrence of symptomatic brain radiation necrosis requiring medical or surgical intervention and confirmed by pathology | 30 days post index procedure
The number of Grade 4 neutropenia events persisting for longer than 5 days | 30 days post index procedure
The number of grade 4 febrile neutropenia | 30 days post index procedure
The number of grade 4 thrombocytopenia or grade 3 thrombocytopenia with hemorrhage | 30 days post index procedure

SECONDARY OUTCOMES:
Rate of any treatment-related adverse events and treatment-related serious adverse events (not including predefined Limiting Toxicities) from first patient enrolled through study completion. | Enrollment through 6 months post index procedure
Change in post-treatment neurological function as assessed by the National Institute of Health Stroke Scale (NIHSS). | Enrollment through 6 months post index procedure
  The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
Change in post-treatment neurological function as assessed by the modified Rankin Scale (mRS). | Enrollment through 6 months post index procedure
  The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability on a scale from 0 (no symptoms at all) to 6 (death).
Technical Success/Feasibility of TheraSphere GBM - ability to deliver the projected radiation absorbed dose (+/- 20%) to the perfused volume for all patients treated with the device. Assessed from pre-screening through post-device delivery PET-CT/MRI. | Pre-screening through post-device delivery PET-CT/MRI.
Objective Response Rate* (ORR) from first patient enrolled through study completion | Enrollment through 6 months post index procedure
Progression Free Survival* (PFS) from first patient enrolled through study completion | Enrollment through 6 months post index procedure
Overall Survival (OS) from first patient enrolled through study completion | Enrollment through 6 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, M.D., Principal Investigator — Northwestern University; Roger Stupp, M.D., Principal Investigator — Northwestern University
Locations (9):
- United States (9):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Mayo Jacksonville, Jacksonville, Florida
  - Northwestern Univerity, Chicago, Illinois
  - Johns Hopkins Interventional Radiology Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Lenox Hill Hospital, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meiselman S, Thomas MA, Giardina JD, Zheleznyak A, Thorek DLJ, Malone CD. Advances in Radioembolization for Liver Cancer. J Vasc Interv Radiol. 2025 Dec;36(12):1876-1881. doi: 10.1016/j.jvir.2025.07.018. PMID 41276366